CLINICAL TRIAL: NCT00341900
Title: Study of Markers of Cosmic Radiation Exposure and Effect Among Flight Crews
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902043; 02-C-N043
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Frequency of Chromosome Aberrations
Keywords: Chromosome Translocations; Cosmic Radiation; Airline Flight Crew; Airlines; Flight Crew; Occupational Exposure
MeSH Terms: conditions — Translocation, Genetic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case: Male pilots with high cosmic radiation exposure

SUMMARY:
Ionizing radiation efficiently induces chromosomal aberrations (CA) and several studies of CA have now been conducted among small groups of flight crews. However, most of the studies only evaluated the unstable aberrations that reflect recent exposures, but not long-term cumulative cosmic radiation exposure. Chromosome painting by fluorescence in situ hybridization (FISH) is a widely used and established cytogenetic method for detecting stable aberrations such as translocations. Thus, FISH can be used for estimating chromosomal damage from cumulative radiation exposure. No large studies of flight crews utilizing FISH have been conducted to date.

We propose a study to measure CA using FISH in a group of pilots estimated to have high comic radiation exposure based on flight histories, i.e., those with long duration flying international routes, and a comparison group of university faculty with minimal flying history. These measurements will be used to determine if pilots have elevated frequencies of CA (specifically stable translocations) as compared with the university faculty. In addition, the frequencies of CA will be examined in relation to the cumulative cosmic radiation dose to determine if there is a dose-response relationship. Individual cumulative doses will be calculated from pilot flight histories using a computer program developed by the FAA which estimates cosmic radiation does by accounting for changes in altitude and latitude, and the 11-year solar cycle at the time of the flight. We will collect information on age, lifestyle factors, diet, health history, family cancer history, and medical radiation exposures from personal interview and self-administered dietary questionaire. These factors may affect the CA frequency and so we plan to adjust for them in the statistical analyses.

Pilots will be identified based on the Allied Pilots Association roster and faculty from a commercial company that maintains a database of university faculty, including those in the Chicago area. Potential participants will be notified of the study by mail and recruited/screened for eligibility over the telephone. We will compensate participants $100 for their time. A field station will be set up at a medical or health clinic convenient to the participants, where interviews Will be conducted and a peripheral blood sample collected. Participants will be notified of the overall study results and may request their personal CA results at the end of the study. Participants may also choose to have additional blood drawn, however this blood sample will be anonymized so that it cannot be linked back to the participant. Genotypic variants in DNA repair (and possibly other) genes will be evaluated for an effect on CA frequency.

DETAILED DESCRIPTION:
Ionizing radiation efficiently induces chromosomal aberrations (CA) and several studies of CA have now been conducted among small groups of flight crews. However, most of the studies only evaluated the unstable aberrations that reflect recent exposures, but not long-term cumulative cosmic radiation exposure. Chromosome painting by fluorescence in situ hybridization (FISH) is a widely used and established cytogenetic method for detecting stable aberrations such as translocations. Thus, FISH can be used for estimating chromosomal damage from cumulative radiation exposure. No large studies of flight crews utilizing FISH have been conducted to date.

In collaboration with the National Institute for Occupational Safety and Health (NIOSH), we proposed a study to measure CA using FISH in a group of pilots estimated to have high comic radiation exposure based on flight histories, i.e., those with long duration flying international routes, and a comparison group of university faculty with minimal flying history. These measurements will be used to determine if pilots have elevated frequencies of CA (specifically stable translocations) as compared with the university faculty. In addition, the frequencies of CA will be examined in relation to the cumulative cosmic radiation dose to determine if there is a dose-response relationship. Individual cumulative doses will be calculated from pilot flight histories using a computer program developed by the FAA which estimates cosmic radiation does by accounting for changes in altitude and latitude, and the 11-year solar cycle at the time of the flight. We will collect information on age, lifestyle factors, diet, health history, family cancer history, and medical radiation exposures from a self-administered study and dietary questionnaire. These factors may affect the CA frequency and so we plan to adjust for them in the statistical analyses.

Pilots were identified based on the Allied Pilots Association roster and faculty from a commercial company that maintains a database of university faculty, including those in the Chicago area. Potential participants will be notified of the study by mail and recruited/screened for eligibility over the telephone. We compensated participants $100 for their time and inconvenience. Two field stations were arranged at the O'Hare UIC medical clinic for pilots and at the UIC Health Services clinic (on campus) for the faculty, where interviews were conducted and a peripheral blood sample collected. Participants will be notified of the overall study results and may request their personal CA results at the end of the study. Participants may also choose to have additional blood drawn, however this blood sample will be anonymized so that it cannot be linked back to the participant. Genotypic variants in DNA repair (and possibly other) genes will be evaluated for an effect on CA frequency.

ELIGIBILITY:
* INCLUSION CRITERIA:

PILOTS:

Subjects will be Chicago based pilots who fly international flights out of Chicago.

Subjects must have worked at least 10 years as an international pilot.

EXTERNAL COMPARISON GROUP:

Subjects must be currently employed as university faculty from the Chicago area.

Pilots and External Comparison Group Subjects:

Age 35-54.

Non-Smoker (less than 100 lifetime cigarettes).

Male.

EXCLUSION CRITERIA:

PILOTS AND EXTERNAL COMPARISON GROUP SUBJECTS:

No personal history of cancer.

No history of chemotherapy.

No history of major diagnostic radiation therapy (e.g., radio-imaging that exposed the large bones or lymph nodes except for routine medical and dental x-rays).

No family history of hereditary diseases (ataxia telangiectasia, Fanconi's anemia, Bloom's syndrome, and xeroderma pigmentosum).

EXTERNAL COMPARISON GROUP SUBJECTS:

Must not have a history of excessive past air travel (defined as no more than an average of one international flight/year and one domestic flight/month).

No history of major illnesses, such as heart disease and diabetes.

Must not have been employed in a clinical or laboratory area that involves exposure to radiation and chemotherapeutic drugs.

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pilots estimated to have high comic radiation exposure based on flight histories.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2001-11-09 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Chromosome translocation frequency | One time point
  Chromosome translocation frequency

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Little, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institute for Occupational Safety and Health, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Yong LC, Sigurdson AJ, Ward EM, Waters MA, Whelan EA, Petersen MR, Bhatti P, Ramsey MJ, Ron E, Tucker JD. Increased frequency of chromosome translocations in airline pilots with long-term flying experience. Occup Environ Med. 2009 Jan;66(1):56-62. doi: 10.1136/oem.2008.038901. Epub 2008 Dec 11. PMID 19074211
- [Background] Grajewski B, Waters MA, Yong LC, Tseng CY, Zivkovich Z, Cassinelli RT 2nd. Airline pilot cosmic radiation and circadian disruption exposure assessment from logbooks and company records. Ann Occup Hyg. 2011 Jun;55(5):465-75. doi: 10.1093/annhyg/mer024. Epub 2011 May 24. PMID 21610083
- [Background] Yong LC, Petersen MR, Sigurdson AJ, Sampson LA, Ward EM. High dietary antioxidant intakes are associated with decreased chromosome translocation frequency in airline pilots. Am J Clin Nutr. 2009 Nov;90(5):1402-10. doi: 10.3945/ajcn.2009.28207. Epub 2009 Sep 30. PMID 19793852